CLINICAL TRIAL: NCT05607472
Title: Factors Associated With Hospitalization for Dengue and Dengue Severity: Hospital-based Cohort Study on Reunion Island
Acronym: DENGUE-RUN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/CHU/37
Record Dates: First submitted 2022-01-06; First posted 2022-11-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Dengue Fever With Warning Signs
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patient with Dengue prognostic purpose (Other): blood samples for bio collection clinical exam : Fitzpatrick phototype classification , Charlson comorbidity classification questionaries : SHERE and EHAD (emotional evaluation), SF-12, EQ-5D-5L, MFIS-5 (Fatigue evaluation)
  Interventions: Other: blood sampling; Other: questionnary of health estate during 18 month

INTERVENTIONS:
Other: blood sampling — blood samples for bio collection
Other: questionnary of health estate during 18 month — clinical exam Charlson comorbidity classification questionaries : SHERE and EHAD (emotional evaluation), SF-12, EQ-5D-5L, MFIS-5 (Fatigue evaluation) during 18 months

SUMMARY:
In recent years, dengue has become endemic on La Réunion island, which has led to subsequent increase of secondary dengue infections, higher severity and higher mortality of the cases referred to the hospital.

This project will investigate the factors associated with the hospitalization for dengue and the factors associated with dengue severity in a hospital-based cohort study conducted over two dengue seasons, as well as the long-term outcomes over aN18-month follow-up.

DETAILED DESCRIPTION:
Dengue is a re-emerging infectious disease caused by the four serotypes of dengue virus, a flavivirus transmitted through the bite of a female Aedes mosquito. Dengue heterotypic cross-immunity (against the four serotypes) is short-lived while dengue homotypic immunity (against one serotype) is supposed to be lifelong allowing the possibility of four dengue episodes in a lifetime. In recent years, dengue has become endemic on Réunion island, which has led to the circulation of multiple serotypes (DEN2 in 2018-2019 and DEN1 in 2020-2021), subsequent increase of secondary dengue infections, higher severity and higher mortality of cases referred to the hospital. This project will investigate both the factors associated with the hospitalization for dengue and the factors associated with dengue severity in a hospital-based cohort study conducted over two dengue seasons, as well as the long-term outcomes over an 18-month follow-up. The investigators hypothesize that in an epidemiological context of endemization (which means in the transition from sporadicity towards endemicity), primary dengue infections will be still prominent and severe dengue will be associated with comorbidities rather to prior infections occurring in healthy backgrounds. The data collection will consist in clinical, biological and survey data. Electronic case report forms will be informed by medical doctors and research assistants in outpatient clinics, emergency departments, intensive care units and short-stay admission units. A biobank will be set up on this occasion including serum, plasma, PBMC, DNA, RNA urine samples and possibly CSF.

The follow-up will screen post-infectious long-term manifestations such as chronic fatigue syndrome, musculoskeletal disorders, anxiodepressive or cognitive disorders, and sequelae 3 months, 6 months 12 months and 18 months after the dengue event.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (including pregnant women) or children (> 8 kg)

* Admitted to the Emergency Department, in the hospital wards, or in outpatient clinics from the two teaching hospitals of Réunion island
* with a definite or probable diagnosis of dengue, as defined by a positive PCR (plasma or urine), NS1 antigen within the first five days of onset of symptoms; or 2 serologies indicating a recent primary or a secondary infection (positive IgM twice or IgG seroconversion x 4 at a minimum of 10 days apart)
* affiliated to a social insurance

Exclusion Criteria:

* refusal of participation as expressed by the patient or its entourage (if the patient is physically unable to give his opinion)
* absence of social insurance

Min Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The relative risk for hospitalization with dengue of any risk factors measured at inclusion ) | 18 months
  The incidence rate ratio (relative risk) for hospitalization with dengue of any risk factors measured at inclusion (first consultation) as identified from a multivariate Poisson regression model for dichotomous outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Manuella POTHIN, Study Director — CHU La Réunion
Locations (1):
- Patrick GERARDIN, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: Undecided